CLINICAL TRIAL: NCT03172273
Title: Early Use of Transjugular Intrahepatic Portosystemic Shunt（TIPS）With Polytetrafluoroethylene(PTFE) Covered Stents in Cirrhotic Patients With Refractory Ascites
Brief Title: Early Use of TIPS With Polytetrafluoroethylene(PTFE) Covered Stents in Cirrhotic Patients With Refractory Ascites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, PhD&MD, Xi'an International Medical Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA-TIPS
Record Dates: First submitted 2017-05-27; First posted 2017-06-01 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Liver Cirrhoses
Keywords: Liver Cirrhosis; Transjugular Intrahepatic Portosystemic shunt; Refractory ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS with PTFE (Experimental): Transjugular Intrahepatic portosystemic shunt with PTFE covered stents
  Interventions: Procedure: TIPS
- paracentesis (Active Comparator): Paracentesis with albumine invision
  Interventions: Procedure: paracentesis

INTERVENTIONS:
Procedure: TIPS — Transjugular intrahepatic portosystemic shunt with covered PTFE
  Arms: TIPS with PTFE
Procedure: paracentesis — paracentasis plus albumine invision
  Arms: paracentesis

SUMMARY:
This multicenter RCT is designed to investigate if TIPS with covered stents improves transplant-free survival for cirrhotic patients with early stage of refractory ascites compared to LVP+albumin during 1 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of liver cirrhosis
* Recurrent and refractory ascites
* Patients with an age between 18 and 65 years old
* Child-Pugh ≤12
* Absence of hepatic encephalopathy
* Patient is willing and able to comply with all study protocol requirements, including specified follow-up and testing.
* Patient, or legal authorized representative, is willing to provide written informed consent prior to enrollment in the study

Exclusion Criteria:

* With more than 6 paracenteses within the last 3 months
* patients expected to receive transplants within the next 6 months or on waiting list
* Usual contra-indication for TIPS: congestive heart failure NYHA>III or medical history of pulmonary hypertension, portal vein thrombosis（>50%）, hepatic polycystosis, intra-hepatic bile ducts dilatation
* Patient has had previous TIPS placement
* Severe liver dysfunction by: Prothrombin index < 40% or total bilirubin > 50μmol/l
* Serum creatinine >133μmol/l
* Severe hyponatremia <125mmol / L
* Uncontrolled sepsis
* Gastrointestinal hemorrhage within 6 weeks of randomization
* Known allergy to albumin
* Pregnant or breast feeding women
* Refusal to participate or patient unable to receive informations or to sign written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival | 12 months

SECONDARY OUTCOMES:
Frequency of paracentesis | 12 months
Frequency of overt Hepatic Encephalopathy | 12 months
  Number of episodes of West Haven grade 2 or greater without precipitating factor
Nutritional status | 12 months
Quality of life | 12 months
Other Liver Disease Complications (Adverse Events) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD&MD, Principal Investigator — Xi'an International Medical Center Hospital
Locations (2):
- China (2):
  - the First Affiliated Hospital, Air Force Medical University, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi

REFERENCES:
- [Background] Bureau C, Thabut D, Oberti F, Dharancy S, Carbonell N, Bouvier A, Mathurin P, Otal P, Cabarrou P, Peron JM, Vinel JP. Transjugular Intrahepatic Portosystemic Shunts With Covered Stents Increase Transplant-Free Survival of Patients With Cirrhosis and Recurrent Ascites. Gastroenterology. 2017 Jan;152(1):157-163. doi: 10.1053/j.gastro.2016.09.016. Epub 2016 Sep 20. PMID 27663604
- [Background] Bai M, Qi XS, Yang ZP, Yang M, Fan DM, Han GH. TIPS improves liver transplantation-free survival in cirrhotic patients with refractory ascites: an updated meta-analysis. World J Gastroenterol. 2014 Mar 14;20(10):2704-14. doi: 10.3748/wjg.v20.i10.2704. PMID 24627607